CLINICAL TRIAL: NCT00659191
Title: A Double-Blind, Parallel, Randomized, Placebo-Controlled, Single and Repeat Dose Escalation First Time in Human Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK1265744 in Healthy Male and Female Subjects and Subjects Infected With HIV
Brief Title: A Healthy Volunteer And Patient Study To Assess The Safety, Tolerability And Pharmacokinetics Of GSK1265744
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111451
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: HIV Infection
Keywords: Healthy volunteer,; HIV infected subjects
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir

INTERVENTIONS:
Drug: GSK1265744

SUMMARY:
This study is a Phase I single and repeat dose escalation study of GSK1265744 in healthy subjects and a single repeat dose cohort in HIV-1 infected subjects. The study is planned to consist of three parts. Part A will enroll two cohorts with a total of 18 subjects in a single dose escalation to evaluate safety, tolerability and PK. Part B plans to enroll three cohorts of 10 subjects to evaluate repeat doses of GSK126744 on safety, tolerability and PK. Part A and B will enroll healthy volunteers. Part C will enroll HIV-1 patients in a single cohort of 10 subjects. This cohort will evaluate the effects of repeat dose on safety, tolerability, PK and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Parts A and B: The subject is healthy. Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and 12-lead ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 55 years of age.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who:

  - Is pre-menopausal with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy, or Is post-menopausal defined as 12 months of spontaneous amenorrhea. A follicle stimulating hormone (FSH) level will be performed to confirm a post-menopausal status. For this study, FSH levels > 40 mlU/ml is confirmatory.
* A male is eligible to enter and participate in the study if he is surgically sterile OR if he either agrees to abstain from sexual intercourse with a female partner or agrees to use a condom/spermicide, in addition to having his female partner use another form of contraception as in protocol
* Body weight >/ 50 kg (110 lbs.) for men and >/ 45 kg (99 lbs) for women and body mass index (BMI) within the range 18.5-31.0 kg/m2 (inclusive).
* A signed and dated written informed consent is obtained from the subject or the subject's legal representative prior to screening.
* Subject must be capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Part C: HIV-infected cohort only: CD4 cell count >/ 200 cells/mm3 and plasma HIV-1 RNA >/ 5,000 copies/mL.
* Part C: HIV-infected cohort only: A pre-baseline viral load measurement will be obtained 7-14 days after the screening visit. The pre-baseline viral load must be within 0.7 log of the screening HIV-1 RNA and must meet the screening HIV-1 RNA (i.e., > 5000) requirements for the subject to be included.

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* Has a positive pre-study Hepatitis B surface antigen; positive hepatitis C (HCV) antibody or detectable HCV ribonucleic acid (RNA); or positive HIV-1 antibody result. NOTE that a positive HIV-1 antibody result is acceptable for those entering the study as a subject infected with HIV-1 (Part C)
* Has a history of regular alcohol consumption averaging >7 drinks/week for women or >14 drinks/week for men within 6 months of the screening visit.

Note: 1 drink is equivalent to 12 g alcohol = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.

* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* The subject has received an investigational drug or participated in any other research trial within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Participation in the study would result in donation of blood in excess of 500 mL within a 56 day period.

Note: This does not include plasma donation.

• History or presence of allergy or intolerance to the study drug or its components or drugs of its class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.

Note: "Study" or "investigational" drugs include GSK1265744 or placebo.

* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* Exclusion criteria for screening ECG as outlined in protocol.

  * Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization).
  * Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], WPW syndrome).
  * Sinus Pauses > 3 seconds.
  * Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject.
  * Non-sustained or sustained ventricular tachycardia (>/3 consecutive ventricular ectopic beats).
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting surgery or percutaneous transluminal coronary angioplasty or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease.
* Has a history of regular use of tobacco- or nicotine-containing products within 3 months of the screening visit.
* The subject has a positive pre-study drug and/or alcohol screen.
* Use of prescription or non-prescription drugs, including antacids, vitamins, herbal and dietary supplements (including St John's Wort and iron supplements) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin values greater than the upper limit of normal. A single repeat is allowed for eligibility determination.
* History of significant renal or hepatic diseases.
* Exclusion Criteria for 24-Hour Screening Holter:

  * Any symptomatic arrhythmia (except isolated extra systoles).
  * Sustained cardiac arrhythmias (such as atrial fibrillation or flutter, supraventricular tachycardia (>/10 consecutive beats), complete heart block).
  * Non-sustained or sustained ventricular tachycardia (defined as >/ 3 consecutive ventricular ectopic beats).
  * Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular (AV) block [2nd degree or higher], WPW syndrome etc.).
  * Sinus Pauses > 3 seconds.
  * 300 or more supraventricular ectopic beats in 24 hours.
  * 250 or more ventricular ectopic beats in 24 hours.

An HIV-infected subject will not be eligible for inclusion in this study if any of the following criteria apply:

* An active Center for Disease Control (CDC) Category C disease [see Appendix 6], except cutaneous Kaposi's sarcoma not requiring systemic therapy during the trial.
* Prior treatment with an integrase inhibitor (>/ 1 dose).
* Serum alanine aminotransferase (ALT) >2 times the upper limit of normal at screening. A single repeat is allowed for eligibility determination.
* Absolute neutrophil counts <1000/uL, hemoglobin <10 g/dL, platelet count <50,000/uL or creatinine clearance <50 mL/minute. A single repeat is allowed for eligibility determination.
* History of clinically relevant pancreatitis or hepatitis within the previous 6 months.
* Treatment with radiation therapy or cytotoxic chemotherapeutic agents within 30 days of study drug administration or anticipated need for such treatment within the study.
* Treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, interferons) or any agent with known anti-HIV activity (such as hydroxyurea or foscarnet) within 30 days of study drug administration
* Treatment with any vaccine within 30 days prior to receiving study medication.
* The subject has a positive pre-study drug screen including amphetamines, barbiturates, cocaine, or PCP.
* Use of multivitamins or antacids within 7 days prior to the first dose of investigational product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Safety evaluations (labs, ECG, blood pressure), and blood sampling for PK, Continuous AE monitoring through study conclusion and follow up, 7-14 days after last dose. For Part C only: anti-viral activity through study conclusion and follow-up. | through study conclusion and follow up, 7-14 days after last dose

SECONDARY OUTCOMES:
GSK1265744 blood levels to determine PK parameters | on days 1 through day 10
Plasma HIV-1 RNA levels | from baseline and at intervals to Day 21
To assess the development of genotypic viral resistance, if appropriate, in HIV cohort.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Madison, Wisconsin